CLINICAL TRIAL: NCT06914869
Title: A Phase I, Randomized, Open-label, Drug-drug Interaction Study to Assess the Effect of Multiple Doses of a Moderate and a Strong CYP3A Inducer on the Pharmacokinetics and Safety of Mavorixafor in Healthy Male and Female Participants
Brief Title: Drug-Drug Interaction Potential of Mavorixafor
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: X4 Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: X4P-001-004
Record Dates: First submitted 2025-02-27; First posted 2025-04-06 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Healthy Participants
MeSH Terms: interventions — mavorixafor; Carbamazepine; efavirenz

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1: Mavorixafor and Carbamazepine (Experimental): Participants will receive a single dose of mavorixafor administered on Day 1 and a single dose of mavorixafor administered on Day 18 on an empty stomach, after an overnight fast (at least 10 hours). Participants will receive carbamazepine administered orally twice daily (BID) on Days 6 through Day 22, 30 minutes after the end of a meal.
  Interventions: Drug: Mavorixafor; Drug: Carbamazepine
- Cohort 2: Mavorixafor and Efavirenz (Experimental): Participants will receive a single dose of mavorixafor administered on Day 1 and a single dose of mavorixafor administered on Day 18 on an empty stomach, after an overnight fast (at least 10 hours). Participants will receive efavirenz administered once daily (QD) on Days 6 through 22, at bedtime, at least 4 hours after the end of a meal.
  Interventions: Drug: Mavorixafor; Drug: Efavirenz

INTERVENTIONS:
Drug: Mavorixafor — Mavorixafor will be administered per schedule specified in the arm description.
Drug: Carbamazepine — Carbamazepine will be administered per schedule specified in the arm description.
  Arms: Cohort 1: Mavorixafor and Carbamazepine
Drug: Efavirenz — Efavirenz will be administered per schedule specified in the arm description.
  Arms: Cohort 2: Mavorixafor and Efavirenz

SUMMARY:
The main purpose of this study is to evaluate drug-drug interaction (DDI) of orally administered mavorixafor with cytochrome P3A (CYP3A) inducers carbamazepine (a strong CYP3A inducer) or efavirenz (a moderate CYP3A inducer) in healthy male and female participants.

ELIGIBILITY:
Key Inclusion Criteria:

* Body mass index (BMI) between 18.5 and 32 kilograms (kg)/square meter (m^2), inclusive, and body weight not less than 50 kg at Screening.
* Nonsmokers (or other tobacco or nicotine-containing products, in any form, including e-cigarettes and vaping) as determined by history (no nicotine use for 6 months before Screening) and by negative cotinine test at Screening and Admission.
* Healthy, determined by prestudy medical evaluation (medical history, physical examination, vital signs, 12-lead electrocardiogram [ECG], and clinical laboratory evaluations) at Screening and Admission. A repeat test (only once per visit) for vitals, ECG, and/or clinical laboratory evaluations may be performed at the investigator's discretion to confirm results.

Key Exclusion Criteria:

* Participant has used an investigational drug (including mavorixafor) within 30 days (90 days for biologics), or 5 half-lives, whichever is longer prior to Screening.
* Participant has a history of or currently suffers from an active illness considered to be clinically significant (CS) by the investigator or any other illness that the investigator considers should exclude the participant from the study or that could interfere with the interpretation of the study results.
* Participant has CS history or evidence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, neurological, immunological, metabolic, allergic, hematological, or psychiatric disorder(s) as determined by the investigator or designee.
* Female participant is breastfeeding, pregnant, or plans to be pregnant within the duration of the study and up to 4 weeks after completion of the study.
* Use any drugs of abuse (medical or recreational) for at least 30 days prior to first study intervention administration as documented by a history and positive results for urine drug screening (for example, cocaine, amphetamines, barbiturates, opiates, benzodiazepines, cannabinoids), at Screening and/or Admission.
* Participant has positive coronavirus disease 2019 test on Admission confirmed by rapid antigen testing.
* Receipt of any vaccine within 30 days prior to first study intervention or plans to receive any vaccination during the study.
* Any other reason that, in the opinion of the investigator, would render the participant unsuitable for study enrollment.

Specific exclusion criteria for Cohort 1:

* Participant with a history of drug-induced bone marrow depression, hepatic disorders (including porphyrias), severe cutaneous reactions, myotonic dystrophy, psychiatric disorders (including psychosis, depression, and suicidal behavior or ideation), epileptic seizures, increased ocular pressure, or urinary retention syndrome.
* Participants with the human leukocyte antigens (HLA)-A*31:01 or HLA-B*15:02 allele, known hypersensitivity, or intolerance to study interventions.
* Participant with sodium/leukocyte/thrombocyte count below the lower limit of normal at Screening and Admission.
* Participant who previously experienced hypersensitivity reaction to anticonvulsants including phenytoin, primidone, and phenobarbital.

Specific exclusion criteria for Cohort 2:

* Participants with previously demonstrated CS hypersensitivity (for example, Stevens-Johnson syndrome, erythema multiforme, or toxic skin eruptions) to efavirenz.
* Participants with a history of serious psychiatric events such as severe depression, suicidal ideation, nonfatal suicide attempts, paranoid and manic reactions.

NOTE: Other protocol-defined inclusion and exclusion criteria may apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2025-02-18 (Actual); Primary Completion 2025-05-19 (Actual); Study Completion 2025-05-19 (Actual)

PRIMARY OUTCOMES:
Cohort 1: Maximum Observed Plasma Concentration (Cmax) of Mavorixafor Without (Day 1) and With (Day 18) Coadministration With Carbamazepine | Predose up to 120 hours postdose on Days 1 and 18
Cohort 1: Area Under the Concentration-time Curve From Time Zero to the Last Quantifiable Concentration (AUC0-last) of Mavorixafor Without (Day 1) and With (Day 18) Coadministration With Carbamazepine | Predose up to 120 hours postdose on Days 1 and 18
Cohort 2: Cmax of Mavorixafor Without (Day 1) and With (Day 18) Coadministration With Efavirenz | Predose up to 120 hours postdose on Days 1 and 18
Cohort 2: AUC0-last of Mavorixafor Without (Day 1) and With (Day 18) Coadministration With Efavirenz | Predose up to 120 hours postdose on Days 1 and 18

SECONDARY OUTCOMES:
Cohort 1: Time to Reach Cmax (Tmax) of Mavorixafor Without (Day 1) and With (Day 18) Coadministration With Carbamazepine | Predose up to 120 hours postdose on Days 1 and 18
Cohort 2: Tmax Mavorixafor Without (Day 1) and With (Day 18) Coadministration With Efavirenz | Predose up to 120 hours postdose on Days 1 and 18
Cohort 1: Predose Concentration (Ctrough) of Carbamazepine | Predose on Days 14, 16, and 18
Cohort 2: Ctrough of Efavirenz | Predose on Days 14, 16, and 18
Cohorts 1 and 2: Number of Participants With Treatment-emergent Adverse Events (TEAEs) | Day 1 up to Day 33

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, Study Director — X4 Pharmaceuticals, Inc.
Locations (1):
- Parexel International LLC, Baltimore, Maryland, United States